CLINICAL TRIAL: NCT04845581
Title: Comparison of the Effectiveness of the Ultrasonic Method and Cone-beam Computed Tomography Combined With Intraoral Scanning and Prosthetic-driven Implant Planning Method in Determing the Gingival Phenotype in the Healthy Periodontium.
Brief Title: Comparison of the Effectiveness of the USG and CBCT Combined With Intraoral Scanning Determing the Gingival Phenotype in the Healthy Periodontium
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: kb245/2018(2)
Record Dates: First submitted 2021-03-22; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-01

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Diagnostic tests: Determination of the gingival phenotype, measure gingival thickness and width of keratinized tissue — Gingival thickness was measured using UGTM method and CBCT/ CAD with PDIP technology at upper incisors and canines in three points localized midbucally : Free gingival thickness (FGT), supracrestal ( SGT) and crestal (CGT). Width of keratinized tissue was measured using periodontal probe calibrated for 1 mm. The gingival phenotype was determined by both methods according to the following criteria: GT ≤ 0,7 mm - thin gingival phenotype, GT > 0,7 mm ≤ 1,0 mm - medium gingival phenotype, GT > 1,0 mm - thick gingival phenotype. Toincrease the repeatability of the results, two researchers tested the same values twice on 2days interval between sessions.

SUMMARY:
Compare two diagnostic methods: UGTM and CBCT/CAD/PDIP in determing the gingival phenotype in group of 30 periodontally healthy patients. Both methods were useful to establishing the gingival phenotype, however, ultrasonic method was more precisely for measurement of gingival thickness. There was positive correlation between the mean values of SGT and WKT and this indicates the need to measure these parameters in order to determine gingival phenotype.

DETAILED DESCRIPTION:
Gingival phenotype (GP) should be determine in each dento-gingival unit as a 3D volume of gingiva with the following parameters: width of keratinized tissue (WKT) and gingival thickness (GT). The phenotype determination is extremely important during many dental procedures, such as in dental surgery, orthodontics, prosthetics or implantology because it allows to dental treatment planning and reduce the risk of complications. Previous methods of determining the gingival phenotype were based on the shape of the crowns of the upper incisors and transparency of the free gingiva. These methods are non-invasive, but innacurate. The gingival phenotype may be determined more precisely by using biometry of WKT and GT. There are several possible methods to measure the thickness of the gingiva, such as bone sounding, cone beam comuted tomography (CBCT) measurement or parallel profile radiographs, CBCT/CAD (CBCT and computer-aided design) and ultrasound method. The ultrasonic gingival tissue measurement (UGTM) method is non-invasive, removes the need for anesthesia, which may increases the volume of tissues, but requires the experience of the researcher. However, it is considered as effective and reproducible method of the measurement soft tissue thickness. CBCT/CAD/PDIP (CBCT/CAD and prosthetic-driven implant planning) method also can be used to establishing the gingival phenotype.

Measurements of WKT are most often carried out using a periodontal probe calibrated every 1mm. In each case, a necessary condition for the proper examination of the patient and determination of GP is healthy periodontium.

ELIGIBILITY:
Inclusion Criteria:

* lack of general diseases
* good oral hygiene
* healthy periodontium - API ratio<15%, BOP<10%
* no loss of clinical attachment in the examined areas (CAL=0)
* no use of drugs
* no addictions, especially cigarette smoking
* no use of mobile prosthetic restorations and orthodontic appliances
* no contraindications for X-ray examinations

Exclusion Criteria:

* general diseases
* poor oral hygiene
* non healthy periodontium - API ratio>15%, BOP>10%
* loss of clinical attachment in the examined areas (CAL>1)
* use of drugs that could influence the structure of the periodontal tissues
* addictions, especially nicotinism
* use of mobile prosthetic restorations and orthodontic appliances
* contraindications for X-ray examinations

Ages: 24 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: male 16 female 14
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Determination the gingival phenotype | october 2018 to august 2019
  The UGTM and CBCT/CAD/PDIP methods are useful to determining of gingival phenotype but more accurate and repeatability is UGTM. The presence of a positive correlation between SGT and WKT indicates the need to measured these parameters for the evaluation of GP. T. It is very important to determine the gingival phenotype for each dento-gingival unit especially before complicated dental treatment.

CONTACTS AND LOCATIONS:
Overall Officials: wojciech bednarz, prof, Study Director — wroclaw medical univeristy
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided